CLINICAL TRIAL: NCT01008839
Title: Protein Synthesis in Midthigh Muscles PET/CT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Thomas Lang, PhD, UCSF
Other Study IDs: Protein Synthesis; TLANG_Protiensynthesis (Registry Identifier: Thomas.Lang PhD Professor in Residence)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Sarcopenia
Keywords: study sarcopenia, which muscle becomes weaker with age
MeSH Terms: conditions — Sarcopenia

GROUPS / COHORTS (2):
- Old age group of healthy women: Old women over 70 years old
- young group of healthy women: aged 25-35 years

SUMMARY:
The purpose of this study is to test a new imaging technique to help scientists study sarcopenia, the process by which muscle becomes weaker with age.

ELIGIBILITY:
Inclusion Criteria:

* young healthy women aged 25-35 years and older healthy women above 70 years old.

Exclusion Criteria:

* no cardiac disease, not taking medication for high blood pressure Asthma HIV any other cardiac conditions

Ages: 25 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy women
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-03